CLINICAL TRIAL: NCT04544605
Title: Special Chinese Medicine Out-patient Programme for Discharged COVID-19 Patients: An Observational Study
Brief Title: Special Chinese Medicine Out-patient Programme for Discharged COVID-19 Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hong Kong Baptist University (Other)
Collaborators: The University of Hong Kong (Other); Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, ZhaoXiang Bian, Chair Professor/Director of Clinical Division, SCM, Hong Kong Baptist University
Other Study IDs: HA Covid-19
Record Dates: First submitted 2020-09-03; First posted 2020-09-10 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Post COVID-19
Keywords: COVID-19; Special Chinese Medicine Out-patient Programme; Discharged COVID-19 Patients Observational Study
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Individualized-Chinese herbal medicine — I. Lung and spleen qi deficiency syndrome Clinical manifestations: shortness of breath, fatigue, fatigue, anorexia, nausea, fullness, weak stool, and uneasiness. The tongue is pale and greasy. Recommended prescription: French Pinellia 9g, Chenpi 10g, Codonopsis 15g, Sunburn Astragalus 30g, Stir-fried Atractylodes 10g, Poria 15g, Huoxiang 10g, Amomum villosum 6g (later), and Licorice 6g
  II. Qi and Yin deficiency syndrome Clinical manifestations: fatigue, shortness of breath, dry mouth, thirst, palpitations, sweating, poor appetite, low or no lever, dry cough and little sputum; dry tongue, fine or weak pulses. Recommended prescription: North and south radix salviae 10g, 15g ophiopogonis, 6g American ginseng, 6g schisandra, 6g gypsum l5g, 10g light bamboo leaves, 10g mulberry leaves, 15g reed root, 15g salviae miltiorrhiza, 6g raw liquorice.

SUMMARY:
According to the ongoing observational studies and the Chinese Medicine practice guideline for COVID-19 patients, the discharged patients with COVID-19 still exhibits certain clinical symptoms such as fatigue, poor appetite, short of breath, palpation, and poor sleep, which could be recognized as two main Patterns in Chinese Medicine, Qi Deficiency of Lung and Spleen and Qi & Yin Deficiency. Based on this, pulmonary rehabilitation to improve lung function upon discharged was proposed. Therefore, even patients with COVID-19 were discharged from hospitals, there are symptoms with significant clinical syndromes in Chinese Medicine perspectives. These symptoms, in terms of syndrome, which could link with the body constitutions, could be due to pre-COVID-19 infection, suffering from infection, or a consequence of post-infection.

This observational study is a rehabilitation programme to elucidate i) whether body constitution is linking with the infection of COVID-19; ii) whether TCM can help the recovery of discharged COVID-19 patients.

DETAILED DESCRIPTION:
This is an observational multi-centered study that will be conducted in the government subsidized tri-partite CM out-patient clinics (Chinese Medicine Clinic cum Training and Research Centres, "CMCTRs").

The study contains two parts as follows:

1. Retrospective Syndrome Survey: Retrospective information will be collected from participants using semi-structured interview and measuring the baseline body constitution before the rehabilitation treatment under the Programme, with the self-developed Body Constitutions Questionnaire.
2. TCM therapeutic assessment: The improvement of clinical symptoms and the status of body constitutions will be periodically evaluated.

Clinical CM Diagnostic Pattern & clinical characteristics assessments, lung function tests, quality of life and no. of western medical consultations will be assessed at each visit for 9 months. Both retrospective and prospective assessments will be done for those participants who have already joined the Rehabilitation Program in CMCTRs.

Sample Size: Estimated at 150 participants.

Treatment of the Rehabilitation Program in CMCTRs:

The treatment is based on individual Chinese Medicine syndrome and clinical symptoms based on the Chinese Medicine practice guideline for COVID-19 patients. Two main Chinese medicine syndromes for patients recovered from COVID-19 with the recommended prescriptions will be included in the Rehabilitation Program.

the participants will receive three months individualized-Chinese herbal medicine treatment in CMCTRs. After the three months treatment, they are free to either continue another three-month treatment or enter into the follow-up period. Each participant will be assessed every month during the treatment and three months after treatment as follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Participants under the COVID-19 Rehabilitation Program who have been previously diagnosed to be infected with COVID-19 and discharged from local hospitals after treatment with western medicine, with negative results from COVID-19 virus detection.

Exclusion Criteria:

* Participants will be excluded if they have one or more of the followings: 1) inability to communicate (e.g. cognitive impairment); 2) history of CHM allergies; 3) incompetent in giving consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients at CMCTRs, previously diagnosed to be infected with COVID-19 and discharged from Hong Kong local hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-09-07 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in CM Diagnostic Pattern & Clinical Characteristics using CM Syndrome Differentiation Assessment | Change from Baseline the CM Diagnostic Pattern & Clinical Characteristics at 9 months
  The changes in participants' health as characterized by CM diagnostic pattern & clinical characteristics using CM Syndrome Differentiation according to the Guidelines for Chinese Medicine New Drug Clinical Study (China Medical Science Press, 2002) will be assessed on each visit during the treatment and follow up period.
Change in Body Constitution Scores using Body Constitution Questionnaires Assessment | Change from Baseline the Body Constitution at 9 months
  The changes in participants' health as characterized by body constitution scores using the Body Constitution Questionnaires for the nine specific types of body constitutions will be assessed on each visit during the treatment and follow up period.

SECONDARY OUTCOMES:
Lung Function Questionnaire in Lung Function Assessment | 9 months
  Lung Function Questionnaire is a simple, brief, self-administered instrument to identify patients appropriate for lung function evaluation by 5 items about the breathing problems &/or frequent cough.
  The questions are:
  1. How often do you cough up mucus?
  2. How often does your chest sound noisy (wheezy, whistling, rattling) when you breathe?
  3. How often do you experience shortness of breath during physical activity (walking up a flight of stairs or walking up an incline without stopping to rest)?
  4. How many years have you smoked?
  5. What is your age?
  Scale:
  For Q1-Q3: 5=Never, 4=Rarely, 3=Sometimes, 2=Often, and 1=Very often For Q4: 5=Never, 4=≦10yrs, 3=11-20yrs, 2=21-30yrs, 1=>30yrs For Q5: 5=<40yrs, 4=40-49yrs, 3=50-59yrs, 2=60-69yrs, 1=≧70yrs
  Score interpretation:
  Total Score of 18 or less suggests increased risk of Chronic Obstructive Pulmonary Disease.
Blood Pressure in 6-minute Walk Test (6MWT) | 9 months
  The six-minute walk test (6MWT) measures the distance the participant is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes. The individual is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway.
  Participant's blood pressure (Systolic/Diastolic) in mmHg will be recorded before and after 6MWT on each visit.
Pulse in 6-minute Walk Test (6MWT) | 9 months
  The six-minute walk test (6MWT) measures the distance the participant is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes. The individual is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway.
  Participant's pulse (beats per minute) will be recorded before and after 6MWT on each visit.
SpO2 in 6-minute Walk Test (6MWT) | 9 months
  The six-minute walk test (6MWT) measures the distance the participant is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes. The individual is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway.
  Participant's SpO2 (%) will be recorded before and after 6MWT on each visit.
Distance Walked in 6-minute Walk Test (6MWT) | 9 months
  The six-minute walk test (6MWT) measures the distance the participant is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes. The individual is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway.
  Participant's distance walked (m) will be recorded during 6MWT on each visit.
Number of Rests in 6-minute Walk Test (6MWT) | 9 months
  The six-minute walk test (6MWT) measures the distance the participant is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes. The individual is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway.
  Participant's number of rests (number) will be recorded during 6MWT on each visit.
MRC Dyspnoea Scale in 6-minute Walk Test (6MWT) | 9 months
  The six-minute walk test (6MWT) measures the distance the participant is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes. The individual is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway.
  Participants' lung function will be assessed using MRC Dyspnoea Scale during 6MWT on each visit, for grading the effect of breathlessness on daily activities. This scale measures perceived respiratory disability and allows the patients to indicate the extent to which their breathlessness affects their mobility.
  The 1-5 grade scale is used alongside the questionnaire to establish the degree of breathlessness related to activity.
Borg Scale of Perceived Exertion in 6-minute Walk Test (6MWT) | 9 months
  The six-minute walk test (6MWT) measures the distance the participant is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes. The individual is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway.
  Participants' Borg Scale of Perceived Exertion ("Borg Score") will be recorded, by asking the participants to rate their exertion on the scale, taking into consideration feelings of physical stress and fatigue focusing on the whole feeling of exertion during 6MWT.
  Scoring used in Borg RPE:
  6=No exertion 7-8=Extremely light 9-10=Very light 11-12=Light 13-14=Somewhat hard 15-16=Hard 17-18=Very hard 19=Extremely hard 20=Maximal exertion
Peak Expiratory Flow (PEF) in Spirometry Assessment | 9 months
  Peak Expiratory Flow (PEF) in litres per second (L/S) is recorded in Spirometry Assessment on each visit to determine participants' lung functionality.
  Peak flow readings are higher when patients are well, and lower when the airways are constricted.
Forced Expiratory Volume in 1 second (FEV1) in Spirometry Assessment | 9 months
  Forced expiratory volume in 1 second (FEV1) in Litres (L) is recorded in Spirometry Assessment on each visit to determine participants' lung functionality by assessing how much air the participants can force from their lungs in one second. Lower FEV-1 readings indicate more significant obstruction.
Force Vital Capacity (FVC) in Spirometry Assessment | 9 months
  Force vital capacity (FVC) in Litres (L) is recorded in Spirometry Assessment on each visit to determine participants' lung functionality by assessing the largest amount of air that the participants can forcefully exhale after breathing in as deeply as they can. A lower than normal FVC reading indicates restricted breathing.
FEV1/FVC ratio (%) in Spirometry Assessment | 9 months
  FEV1 and FVC recorded will be used to calculate the FEV1/FVC ratio (FEV1%) which is the ratio of FEV1 to FVC. In healthy adults this should be approximately 70-80% (declining with age). In obstructive diseases (asthma, COPD, chronic bronchitis, emphysema) FEV1 is diminished because of increased airway resistance to expiratory flow.
  FEV1% of the participants are recorded during each visit, to assess any increased airway resistance to expiratory flow. In restrictive diseases (such as pulmonary fibrosis) the FEV1 and FVC are both reduced proportionally and the value may be normal or even increased as a result of decreased lung compliance.
Quality of Life (WHO-QOL BREF HK) | 9 months
  The World Health Organization Quality of Life Brief Assessment [WHOQOL-BREF (HK)] (Leung, K F; Tay, M., Cheng, S. S. W., Lin, 1997) was validated in Hong Kong and widely use in academia and clinicians since 1997. This is a 5-point Likert scale with a total of 28 Questions to identify the perceived QOL of the participants. There are four domains namely Physical Health, Psychological, Social and Environment domains with a maximum of 100.
Assessment on Western Medicine Visit Frequency | 9 months
  Frequency of clinic/hospital visits for western medicine during the treatment and follow up period

CONTACTS AND LOCATIONS:
Overall Officials: Yi Bin FENG, PhD, Principal Investigator — School of Chinese Medicine, LKS Faculty of Medicine, The University of Hong Kong; Ching LIONG, PhD, Principal Investigator — School of Chinese Medicine, The Chinese University of Hong Kong
Locations (1):
- School of Chinese Medicine, Hong Kong Baptist University, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Undecided